CLINICAL TRIAL: NCT02094495
Title: Pilot Study to Evaluate the Knowledge and Understanding on Tamoxifen Therapy for Breast Cancer Patients
Brief Title: Pilot Study About Tamoxifen Therapy for Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Eun Sook Lee, Chief, Center for Breast Cancer, National Cancer Center, Korea
Other Study IDs: NCC 2014-0112-0001
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: Tamoxifen; Breast cancer; Knowkedge
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- breast cancer group: Taking tamoxifen

SUMMARY:
The aim of this study are to to evaluate the knowledge and understanding on tamoxifen theraphy for breast cancer patients and examine the decision conflict scale and satisfaction with decision scale while making decision to take tamoxifen.

DETAILED DESCRIPTION:
The knowlege questionnaire about tamoxifen was developed by the medication guides that provide for patients taking tamoxifen and hormone therapy for breast cancer fact sheet from National Cancaer Institute. Several experts in the field of breast cancer and gynecologic cancer are going to review and indicate the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* The breast cancer patients who take tamoxifenExclusion Criteria:

Exclusion criteria

* The patients who do not agree to participate in this study
* The paitents who have trouble with understanding and reading Korean.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients who take tamoxifen at National Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The knowledge questionnaire about tamoxifen | The study outcome measure will be assessed by face-to-face, one time.
  There are no more follow up except one time

SECONDARY OUTCOMES:
Decision Conflict Scale | The study outcome measure will be assessed by face-to-face , one time.
  There are no more follow up except one time.

OTHER OUTCOMES:
1. Satisfaction with Decision scale | The study outcome measure will be assessed by face-to-face , one time.
  There are no more follow up except one time
Quality of life (EQ-5D, VAS) | The study outcome measure will be assessed by face-to-face, one time.
Female Sexual Function Index - 6 items, Korean version | The study outcome measure will be assessed by face-to-face, one time.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Sook Lee, MD, PhD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- Center for Breast Cancer, National Cancer Center, Goyang-si, Gyeonggi-do, South Korea